CLINICAL TRIAL: NCT01958346
Title: New Maneuver to Facilitate Fiberoptic Intubation for Difficult Airway: A Prospective, Randomized Study
Brief Title: New Maneuver to Facilitate Fiberoptic Intubation for Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enrico Camporesi (Other)
Responsible Party: Sponsor-Investigator, Enrico Camporesi, Anesthesiologist, University of South Florida
Organization: University of South Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00008289
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Results first posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Anticipated Difficult Airway
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fiberoptic Intubation Alone (Sham Comparator): Intubation with fiberoptic scope assistance
  Interventions: Other: Sham; Device: Fiberoptic Intubation
- Fiberoptic Intubation with lingual traction (Experimental): Intubation with fiberoptic scope assistance and lingual traction maneuver provided by a second anesthesiologist
  Interventions: Other: Lingual Traction; Device: Fiberoptic Intubation

INTERVENTIONS:
Other: Lingual Traction — The tongue pulling maneuver consists of grasping the tongue with 4x4cm gauze and gently pulling the tongue out until resistance is met.
  Arms: Fiberoptic Intubation with lingual traction
Other: Sham — Standard of care fiberoptic intubation without any additional experimental maneuvers
  Arms: Fiberoptic Intubation Alone
Device: Fiberoptic Intubation

SUMMARY:
We propose the additional technique of lingual traction or "tongue pulling" in conjunction with use of the flexible fiberoptic bronchoscope for facilitating successful first attempts at and decreasing time to intubation of the difficult airway and rescuing otherwise failed intubation attempts. Induction of general anesthesia causes relaxation and approximation of the soft palate, base of the tongue, epiglottis, and posterior pharyngeal wall, creating unfavorable anatomic changes in the pharynx for successful intubation. The use of lingual traction can assist in diminishing these problems by clearing the tongue away from the soft palate and uvula and lifting the epiglottis from the posterior pharyngeal wall, especially in the unanticipated difficult airway patient.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* With ASA (American Society of Anesthesiologists) physical status I-III
* With anticipated difficult airway
* Scheduled for elective surgery requiring orotracheal intubation (populations such as elective hip and knee arthroplasty patients)
* Provide written consent

Exclusion Criteria:

* With (American Society of Anesthesiologists) ASA physical status IV
* Pregnant
* Require rapid-sequence induction
* Require a non-standard tracheal tub
* Unable to provide written consent
* At risk for pulmonary aspiration of gastric content

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devanand Mangar, MD, Study Director — Florida Gulf-to-Bay Anesthesiology
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

REFERENCES:
- [Background] Peterson GN, Domino KB, Caplan RA, Posner KL, Lee LA, Cheney FW. Management of the difficult airway: a closed claims analysis. Anesthesiology. 2005 Jul;103(1):33-9. doi: 10.1097/00000542-200507000-00009. PMID 15983454
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Umesh G, George M, Venkateswaran R. Tongue traction is as effective as jaw lift maneuver for Trachlight-guided orotracheal intubation. Acta Anaesthesiol Taiwan. 2010 Sep;48(3):130-5. doi: 10.1016/S1875-4597(10)60044-6. PMID 20864061
- [Background] Rewari V, Ramachandran R, Trikha A. Lingual traction: a useful manoeuvre to lift the epiglottis in a difficult oral fibreoptic intubation. Acta Anaesthesiol Scand. 2009 May;53(5):695-6. doi: 10.1111/j.1399-6576.2009.01934.x. No abstract available. PMID 19419380

RESULTS

PARTICIPANT FLOW:
Groups:
- Fiberoptic Intubation Alone: Sham: Standard of care fiberoptic intubation without any additional experimental maneuvers
  Fiberoptic Intubation
- Fiberoptic Intubation With Lingual Traction: Lingual Traction: The tongue pulling maneuver consists of grasping the tongue with 4x4cm gauze and gently pulling the tongue out until resistance is met.
  Fiberoptic Intubation
Period: Overall Study
Arm/Group | Fiberoptic Intubation Alone | Fiberoptic Intubation With Lingual Traction
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fiberoptic Intubation Alone | Fiberoptic Intubation With Lingual Traction | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.5) | 56.7 (13.9) | 56.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 39 | 39 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 39 | 39 | 78
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Intubations on First Attempt; Grade(s) Were Not Measured.
Time Frame: At Intubation
Measure: Number; unit: participants
Arm/Group | Fiberoptic Intubation Alone | Fiberoptic Intubation With Lingual Traction
Number analyzed (Participants) | 39 | 39
participants | 29 | 36

2. Secondary Outcome: Sore Throat Grade on First Postoperative Day
Description: Patients will be asked to rate their sore throat qualitatively as none, mild, moderate, or severe
Time Frame: Postoperative day one
Measure: Number; unit: participants
Arm/Group | Fiberoptic Intubation Alone | Fiberoptic Intubation With Lingual Traction
Number analyzed (Participants) | 39 | 39
participants | 10 | 14

ADVERSE EVENTS:
Time Frame: Post operative day 1
Description: Sore throats were qualitatively scored by the patient as none, mild, moderate, or severe.
Arm/Group | Fiberoptic Intubation Alone | Fiberoptic Intubation With Lingual Traction
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 3/39 | 6/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fiberoptic Intubation Alone (N=39) | Fiberoptic Intubation With Lingual Traction (N=39)
Sore Throat (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No